CLINICAL TRIAL: NCT05995171
Title: Long Term Outcome of Easophageal Atresia : Transmics Profiles in Adolescence
Acronym: TransEAsome
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022_0483
Record Dates: First submitted 2023-07-31; First posted 2023-08-16 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Atresia
MeSH Terms: conditions — Esophageal Atresia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Esophageal atresia arm: Patient with esophageal atresia
  Interventions: Other: Questionnaire
- control arm: Patient without esophageal atresia
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Quality of life questionnaires will be used specifically for this research: Pediatric Quality of Life Invertory and EA-QoL

SUMMARY:
Oesophageal atresia (OAEA), a malformation of the oesophagus present from birth, is characterized by the interruption of the continuity of the oesophagus, which then ends in a cul-de-sac. (Source: Fimatho) An operation is then required to restore continuity to the esophagus. Although this operation enables the vast majority of children to survive the neonatal period, health problems such as gastro-oesophageal reflux, eating difficulties, respiratory problems and growth problems persist throughout life.

The aim of the project is to create a prospective cohort of adolescents aged 13/14, nested in the national AO registry. of adolescents born with esophageal atresia, including a biobank of esophageal mucosa and plasma blood samples. Once the clinical and omic data have been collected, the data will be transferred to the France Cohortes information system for analysis, in order to assess the long-term outcome of this rare disease and establish multi-omic profiles. Once the clinical data have been collected and the omics data (derived from analysis of the biobank's biological samples) have been generated, they will be analyzed by the project partners to assess the long-term outcome of OA and establish multiomic profiles. The raw data will be available on the France Cohorte platform.

ELIGIBILITY:
Inclusion Criteria:

* For the oesophageal atresia group :
* Born with oesophageal atresia (EA) in France or in French overseas departments and territories
* Anastomosis performed
* Included into the ReNaTo registry
* Aged 13 or 14 during the recruitment period
* Patient willing to comply with all study procedures and duration
* Patient will social security

For the blood sub-study :

* Upper GI endoscopy performed as part of care between 13 and 14 years of age with esophageal mucosal biopsy sampling
* Patient having given written consent to participate in the study

For the control arm:

* Upper GI endoscopy performed as part of care between 10 and 14 years of age with oesophageal mucosal biopsy sampling
* Upper GI endoscopy performed as part of care for chronic or acute digestive signs to rule out organic etiology (peptic esophagitis, gastric esophagitis, eosinophilic esophagitis or ulcer)
* Normal endoscopy and histology
* No chronic progressive disease

Exclusion Criteria:

* For the oesophagal atresia arm :
* Concurrent participation in an interventional trial and in the 3 months prior to inclusion
* Parents refusing to participate in the study

For the control arm :

* Histologically non-normal esophageal biopsy
* Parents refusing to participate in the study
* Child with known organic pathology

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged 13 to 14 born with oesophageal atresia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-11-14 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
prevalence of gastroesophageal reflux disease (GERD) in children born with esophageal atresia | 13-14 years
  GERD = [pH/impedance-metry demonstrating pathological GERD and/or if lesions of peptic esophagitis are observed at an endoscopy in the year preceding the visit or if the child has a history of complicated GERD leading to anti-reflux surgery]

SECONDARY OUTCOMES:
Quality of life, nutritional status and respiratory complications | 13-14 years
  Quality of life= EA-QoL and PedsQL The quality of life of patients in adolescence will be assessed by means of the following quality of life scales at the age of 13-14 years: PedsQL (13) and EA-QoL (11) by both the patient and a parent. Scale scores will be calculated in accordance with the authors' instructions.
  * Nutritional status will be assessed by weight and height, and by calculating the weight/height z-score and BMI z-score using the World Health Organisation growth curves as a reference (14).
  * Frequency of respiratory complications, assessed during clinical examination (hacking cough during infections, chronic cough, asthma, exertional symptoms (cough, dyspnoea), atopy, wheezing and/or stridor/corniness).
Omics and multi omics profiles in plasma | 13-14 years
Factors associated with GERD | Birth,1 year, 6 years and 13-14 years
  It will be determined from patient characteristics at birth, 1 year, 6 years and 13-14 years (ante-natal data, vital signs, presence of associated malformations, type of atresia, surgical procedures performed, surgical/digestive/respiratory/neuro-orthopaedic complications, type of diet and schooling).
Omics and multi omics profiles in esophageal biopsiesfor patient having 1 biopsy | 13-14 years
  metabolites, proteins and methylation
Omics and multi omics profiles in esophageal biopsies for patient having more than 1 biopsy | 13-14 years
  metabolites, proteins and methylation

CONTACTS AND LOCATIONS:
Locations (33):
- France (31):
  - CHU de Lille Hôpital Jeanne de Flandre, Lille, Nord
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - HLC Hôpital Mère Enfant, Bron
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHI Créteil, Créteil
  - CHU Dijon, Dijon
  - CHU Grenoble, La Tronche
  - AP-HP Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHU Le Mans, Le Mans
  - CHU Limoges, Limoges
  - AP-HM Hôpital La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy Hôpital Brabois, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - CHU Orléans, Orléans
  - AP-HP Hôpital Armand Trousseau, Paris
  - AP-HP Hôpital Necker, Paris
  - AP-HP Hôpital Robert Debré, Paris
  - CHU Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
- CHU Fort de France, Fort-de-France, Martinique
- CHU de Saint Denis de la Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leroy M, Aumar M, Duhamel M, Dauchet L, Figeac M, Gaillard S, Hankard R, Labreuche J, Marot G, Reversat J, Armand V, Salzet M, Sfeir R, Vandel J, Gottrand F. Long-term outcome of oesophageal atresia in adolescence (TransEAsome): a national French cohort study protocol. BMJ Open. 2025 Jan 11;15(1):e086303. doi: 10.1136/bmjopen-2024-086303. PMID 39800411